CLINICAL TRIAL: NCT01408459
Title: Adherence Dynamics for Whole Food Interventions in African-American Men
Acronym: DAPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2006-0354
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Prostate cancer prevention
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tomato product (Active Comparator): Motivational telephone counseling weekly
  Interventions: Dietary Supplement: Tomato Product
- Control (Placebo Comparator): No Motivation telephone Counseling
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Tomato Product — Motivational Telephone Counseling weekly
  Other Names: Intervention group
  Arms: Tomato product
Dietary Supplement: Control — No Motivational telephone Counseling
  Other Names: Control Group
  Arms: Control

SUMMARY:
The purposes of this study are to explore the dynamics of adherence, using a simple whole food intervention strategy, both prior to and during the intervention period and to identify nutrient shifts in self-selected diets and to determine health risks (blood pressure, hyperlipidemia, and body weight) that may have resulted from increased tomato product consumption.

DETAILED DESCRIPTION:
African-American (AA) men suffer the greatest proportion of health disparities of any studied category and adherence to advice among this group has been vastly understudied.

Although there are several ongoing trials for behavioral change, either of diet or lifestyle, enrollment rates of AA men (< 25%) often provide insufficient numbers to evaluate adherence issues separately.

Tomatoes, more than lycopene alone, may have beneficial effects on prostate health, including BPH and prostate cancer. Efficacy trials would require long-term adherence to high levels of tomato product (TP) consumption.

ELIGIBILITY:
Inclusion Criteria:

* African-American men aged ≥ 50 yr who recently were found to have serum prostate specific antigen (PSA) concentrations of >2.5 ng/mL with negative prostate biopsy for prostate cancer.
* English literacy
* willing to consume tomato products on a regular basis.

Exclusion Criteria:

* prostate cancer diagnosis
* other cancers < 5 yrs postdiagnosis except for melanoma
* already consuming four 1/2 cup servings of tomato products/wk.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-01-04 (Actual); Primary Completion 2008-08-30 (Actual); Study Completion 2008-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eunyoung Park, M.S., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Park E, Stacewicz-Sapuntzakis M, Sharifi R, Wu Z, Freeman VL, Bowen PE. Diet adherence dynamics and physiological responses to a tomato product whole-food intervention in African-American men. Br J Nutr. 2013 Jun 28;109(12):2219-30. doi: 10.1017/S0007114512004436. Epub 2012 Nov 19. PMID 23200261
- See also: Pubmed — http://www.ncbi.nlm.nih.gov/pubmed/23200261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical Clinic from June 2007 to Aug 2008
Period: Overall Study
Arm/Group | Tomato Product | Control
Started | 22 | 15
Completed | 21 | 14
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tomato Product | Control | Total
Number analyzed (Participants) | 22 | 15 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (7.2) | 68.4 (7.44) | 67.1 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 22 | 15 | 37

OUTCOME MEASURES:

1. Primary Outcome: Tomato Product Intake Between Different Groups
Description: The intervention group: aimed to achieve the goal of more than five servings of TP/week while control group aimed to eat vegetable instead of tomatoes.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: servings/week
Arm/Group | Tomato Product | Control
Number analyzed (Participants) | 22 | 15
servings/week | 6.1 (2.1) | 0.0 (0.0)

2. Secondary Outcome: Diet Adherence to Tomato Product Consumption Between Different Groups
Description: Using 24-hr recall weekly, consumption of tomato product was measured by serving size.
Time Frame: 3 months
Population: Unit: Number of Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Tomato Product | Control
Number analyzed (Participants) | 22 | 15
Participants | 18 | 5

3. Secondary Outcome: Consumption of Tomato Products Between Different Groups
Description: Using 24-hr diet recall, types of tomato products were counted.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Tomato Product | Control
Number analyzed (Participants) | 22 | 15
participants | 22 | 0

4. Secondary Outcome: Differences in Dietary Lycopene Intake Between Different Groups
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Tomato Product | Control
Number analyzed (Participants) | 22 | 15
mg/day | 20.6 (11.3) | 7.25 (9.6)

5. Secondary Outcome: Plasma Lycopene Concentration Between Different Groups
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Tomato Product | Control
Number analyzed (Participants) | 21 | 12
µmol/L | 0.63 (0.4) | 0.41 (0.2)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Tomato Product | Control
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/15
Other Adverse Events (participants affected / at risk) | 0/22 | 0/15

LIMITATIONS AND CAVEATS:
The number of phone calls and collected diet recalls between groups was different because of concern that the control group would increase their tomato product intake.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes